CLINICAL TRIAL: NCT06152237
Title: A Multicenter, Open Label, Randomized, Dose-Escalation and Dose-Expansion Study of the Safety, Tolerability, and Efficacy of a Single Intrathecal Administration of TSHA-102, an AAV9-Delivered Gene Therapy, for the Treatment of Pediatric Females With Rett Syndrome
Brief Title: Safety and Efficacy of TSHA-102 in Pediatric Females With Rett Syndrome (REVEAL Pediatric Study)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Taysha Gene Therapies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TSHA-102-CL-102
Record Dates: First submitted 2023-11-21; First posted 2023-11-30 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Rett Syndrome
Keywords: Rett Syndrome; Neurodevelopmental Disorder; MECP2
MeSH Terms: conditions — Rett Syndrome; Neurodevelopmental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cohort 1 (Experimental): Dose Level 1
  Interventions: Genetic: TSHA-102
- Cohort 2 (Experimental): Dose Level 2
  Interventions: Genetic: TSHA-102

INTERVENTIONS:
Genetic: TSHA-102 — TSHA-102 is a recombinant, non-replicating, self-complementary AAV9 (scAAV9) vector encoding for the miniMECP2 gene. TSHA-102 is a one-time intrathecal (IT) administration.

SUMMARY:
The REVEAL Pediatric Study is a multi-center, Phase 1/2 open-label, dose-escalation and dose-expansion study of TSHA-102, an investigational gene therapy, in pediatric females with Rett Syndrome.

The safety, tolerability, and preliminary efficacy of two dose levels will be evaluated. The study duration is up to 6 years.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a confirmed diagnosis of classical/typical Rett Syndrome with a documented mutation of the MECP2 gene that results in loss of function.
* Participant is between ≥5 to ≤8 years of age at the time of consent.
* Participant must be up to date with all relevant local vaccination requirements, with last vaccination dose received at least 42 days prior to the start of the immunosuppression regimen.
* Participant's parent/caregiver must be willing to allow participant to receive blood or blood products for the treatment of an AE if medically needed.

Exclusion Criteria:

* Participant has another neurodevelopmental disorder independent of the MECP2 gene loss of function mutation, or any other genetic syndrome with a progressive course.
* Participant has a history of brain injury that causes neurological problems.
* Participant had grossly abnormal psychomotor development in the first 6 months of life.
* Participant has a diagnosis of atypical Rett syndrome.
* Participant has an MECP2 mutation that does not cause Rett syndrome.
* Participant requires non-invasive and invasive ventilatory support.
* Participant has contraindications for IT administration of TSHA-102 or lumbar puncture procedure, other medical conditions, or contraindications to any medications required for IT administration.
* Participant has acute or chronic hepatitis B or C infections.

Ages: 5 Years to 8 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2023-12-12 (Actual); Primary Completion 2028-11-02 (Estimated); Study Completion 2031-11-02 (Estimated)

PRIMARY OUTCOMES:
Primary Safety | Baseline through week 52
  The incidence of participants experiencing any treatment-emergent adverse events (AEs) and serious adverse events (SAEs)

SECONDARY OUTCOMES:
Exploratory Efficacy | Baseline through week 52
  Change from baseline in participant's status after TSHA-102 administration as assessed by Clinical Global Impressions Improvement (CGI-I). This 7-point scale (1 = very much improved, 7 = very much worse, etc.) is used by the clinician to assess the participant's overall performance status; higher scores indicate increased severity.
Exploratory Efficacy | Baseline through week 52
  Change from baseline in participant's status after TSHA-102 administration as assessed by Revised Motor Behavior Assessment (R-MBA). This 34-item questionnaire with scores of 0-4 will be administered by a cliniciant to indicate frequency of daily activities (behavioral/social, respiratory, motor/physical, etc.) in participants with Rett Syndrome. Higher scores correlate with greater clinical severity of disease.
Exploratory Efficacy | Baseline through week 52
  Change from baseline in participant's status after TSHA-102 administration as assessed by Rett Syndrome Behavior Questionnaire (RSBQ). The RSBQ is a 45-item questionnaire and is completed by the participant's Caregiver. Scores (0 = not true, 1 = somewhat/sometimes true, or 2 = very true) are applied to subscales including General Mood, Breathing Problems, Fear/Anxiety, Walking/Standing, etc.; higher scores indicate greater severity.
Exploratory Efficacy | Baseline through week 52
  Change from baseline in participant's status after TSHA-102 administration as assessed by Clinical Global Impressions-Severity (CGI-S). This 7-point scale (1 = normal - not I'll all all, 7 = extremely ill, etc.) will be administered by a clinician, based on their experience with patients with the same diagnosis. A higher score indicates greater severity of illness.
Exploratory Efficacy | Baseline through week 52
  Change from baseline in quantitative EEG findings with auditory evoked potential and visual evoked potentials (AEP and VEP). This testing will provide a measure of the electrophysiologic responses of the brain to visual and auditory stimuli.
Exploratory Efficacy | Baseline through week 52
  The percent change from the steroid-free baseline period in monthly countable seizure frequency (MCSF). This testing will provide a measure of participants with seizure freedom following administration of TSHA-102.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Pisani, M.D., Study Director — Taysha Gene Therapies
Locations (5):
- United States (3):
  - Rush University Medical Center & Children's Hospital, Chicago, Illinois
  - Gillette Children's Specialty Healthcare, Saint Paul, Minnesota
  - Washington University, St. Louis, St Louis, Missouri
- CHU Ste-Justine, Montreal, Quebec, Canada
- Children's Neurosciences, Evelina London Children's Hospital, Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No